CLINICAL TRIAL: NCT01713049
Title: Use of 18F-FLT Positron Emission Tomography to Evaluate the Suspicious Findings on Mammography and Breast Ultrasound: A Pilot Study
Brief Title: 18F-FLT PET for Suspicious Findings on Mammography and Breast Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201001043M
Record Dates: First submitted 2012-10-21; First posted 2012-10-24 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2010-08

CONDITIONS: Breast Neoplasms
Keywords: FLT PET; breast neoplasms; mammography; breast ultrasound
MeSH Terms: conditions — Breast Neoplasms | interventions — alovudine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-FLT (Other): 18F-FLT PET for Suspicious Findings on Mammography and Breast Ultrasound.
  Interventions: Drug: 18F-FLT

INTERVENTIONS:
Drug: 18F-FLT — 0.07 mCi/kg of 18F-FDG will be injected intravenously. The data acquisition will be started at 90 minutes after the injection using 2-D acquisition from a GE DISCOVERY ST PET/CT scanner (GE Medical Systems, Milwaukee, WI).
  Other Names: FLT

SUMMARY:
The purpose: To investigate the diagnostic accuracy of 18F-FLT PET for the suspicious lesions on mammograms and ultrasound.

DETAILED DESCRIPTION:
1. To investigate the diagnostic accuracy of 18F-FLT PET for the suspicious lesions on mammograms and ultrasound, using the pathologic result of biopsy as gold standard, and to determine whether 18F-FLT PET can increase the specificity in breast lesion diagnosis and thus reduce the unnecessary biopsy.
2. To evaluate whether 18F-FLT PET is a cost-effective imaging modality for breast cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 20 to 80 years
2. women who have localized findings on mammography and / or ultrasound and will receive biopsy.
3. The lesions on the conventional imaging measure >=1cm
4. WBC count >=3000/L, or platelet>=75,000/L
5. Liver function, AST or ALT < 78 U/L
6. Renal function, Creatinine < 2.0 mg/dl.The laboratory examinations should be performed within 4months before our study.

Exclusion Criteria:

1. Pregnant women or who are planning to be pregnant.
2. Known cancers in other organs.
3. Women who are not able to cooperate with the PET/CT examination.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the diagnostic accuracy of 18F-FLT PET for the suspicious lesions on mammograms and ultrasound, using the pathologic result of biopsy as gold standard. | The biopsy procedures will be scheduled as soon as possible and should be finished within 2 months after 18F-FLT PET.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Wang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Medical Imaging NTUH, Taipei, Taiwan